CLINICAL TRIAL: NCT06767202
Title: Relationship Between Exposure to Phenols and Pregnancy Outcomes After Embryo Transfer
Status: Completed | Type: Observational
Sponsor: keqin liu (Other)
Responsible Party: Sponsor-Investigator, keqin liu, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: liukeqin0208
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Embryo Transfer
Keywords: Embryo Transfer; Dietary polyphenols; bisphenols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women undergoing assisted reproductive technology in Tongji Hospital, Wuhan City, Hubei Pro: 1. Chinese citizens over the age of 20;
  2. IVF/ICSI assisted reproductive treatment in our center;
  3. Complete clinical data, reproductive outcomes and questionnaire data of both sexes;
  4. Knowing about this research and voluntarily accepting this research;

SUMMARY:
The goal of this observational study is to explore the association between phenol exposure and pregnancy outcome after embryo transfer. The main question it aims to answer [is/are]:

Whether exposure to phenols is associated with adverse pregnancy outcomes in pregnant women undergoing assisted reproductive technology?

DETAILED DESCRIPTION:
First of all, paper questionnaires were used in this study, including general information questionnaire, health effect questionnaire, health survey summary form, and dietary assessment questionnaire. Secondly, obtain the relevant information of the medical record system, including: assisted reproduction protocol, IVF examination results, B-ultrasound examination results, laboratory test indicators, pregnancy outcome information and newborn information. Finally, urine samples were detected using a high performance liquid chromatography mass spectrometer.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese citizens over the age of 20;
2. IVF/ICSI assisted reproductive treatment in our center;
3. Complete clinical data, reproductive outcomes and questionnaire data of both sexes;
4. Knowing about this research and voluntarily accepting this research;

Exclusion Criteria:

1. The patient receives sperm or egg donation treatment;
2. The patient gave up the egg collection operation due to various reasons, and the cycle was canceled;
3. The patient abandons treatment before achieving clinical pregnancy, but the fertile frozen embryo is not transferred;
4. There are contraindications to pregnancy, such as serious liver and kidney diseases, malignant tumors, serious mental diseases, uncorrected coagulation function abnormalities or endocrine indicators abnormalities;
5. Incomplete or missing clinical data or follow-up data;

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women undergoing assisted reproductive technology in Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei Province, China from 2024 to 2025
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of clinical pregnancy patients | From the date of randomization until the termination of pregnancy
  Rate of biochemical pregnancy, clinical pregnancy and post-natal patients

SECONDARY OUTCOMES:
Rate of the health newborn | From the date of randomization until the termination of pregnancy
  gestational age/preterm birth, physical health at birth, the incidence of systemic abnormalities or diseases, and other health outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive center，tongji hospital，huazhong university of science and technology, Wuhan, Hubei, China